CLINICAL TRIAL: NCT02130505
Title: Inflammatory Aspects of Glucose in Hyperlipidemia and Diabetes
Acronym: INFORM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Franciscus Gasthuis (Other)
Responsible Party: Principal Investigator, M.A. de Vries, MD, Sint Franciscus Gasthuis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL17100.101.07
Record Dates: First submitted 2014-04-21; First posted 2014-05-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Atherosclerosis; Leukocyte Activation Disorder; Type 2 Diabetes Mellitus; Familial Combined Hyperlipidemia
MeSH Terms: conditions — Atherosclerosis; Diabetes Mellitus, Type 2; Hyperlipidemia, Familial Combined | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- T2DM (Active Comparator): Patients with type 2 diabetes mellitus, defined as having met the diagnostic criteria as outlined by the World Health Organization
  Interventions: Dietary Supplement: OGTT
- FCH (Active Comparator): Patients with familial combined hyperlipidemia, defined as familial hyperlipidemia with a dominant inheritance pattern, elevated plasma apolipoprotein (apo) B concentrations (>1.2 g/L) and elevated triglyceride (TG) levels (>1.7 mmol/L) at the time of diagnosis
  Interventions: Dietary Supplement: OGTT
- FH (Active Comparator): Patients with familial hyperlipidemia, defined as having met the diagnostic criteria as outlined by the world Health Organization
  Interventions: Dietary Supplement: OGTT
- Healthy controls (Active Comparator): Healthy controls
  Interventions: Dietary Supplement: OGTT

INTERVENTIONS:
Dietary Supplement: OGTT — Oral glucose tolerance test (OGTT) with 75 g of oral anhydrous glucose

SUMMARY:
In this study, we will investigate both inflammatory systems in healthy volunteers and patients with T2DM on insulin therapy and hyperlipidemia (both familial hyperlipidemia (FH) and familial combined hyperlipidemia (FCH)) during an OGTT.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is number one killer in the Netherlands. Insulin resistance and dyslipideima are the main causes of CVD. Recently, we have shown that there is an acute leukocyte activation after an oral glucose tolerance test (OGTT) in patients with newly-diagnosed diabets mellitus type 2 (T2DM). Leukocyte activation is an important and obligatory aspect in the process of atherosclerosis. Complement system is another important inflammatory component in atherosclerosis, which becomes activated in the postprandial phase.

In this study, we will investigate both inflammatory systems in healthy volunteers and patients with T2DM on insulin therapy and hyperlipidemia (both familial hyperlipidemia (FH) and familial combined hyperlipidemia (FCH)) during an OGTT.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Aged 45-65 years
* BMI < 35 kg/m2

Exclusion Criteria:

* Emotionally and intellectually not capable to decide about participation in the study and the consequences of participation. Subjects who are not able to understand the patient information
* Diabetes mellitus treated with oral antidiabetic medicine
* Type 1 diabetes mellitus
* Peripheral artery and/or coronary disease
* Untreated hypertension
* Alcohol use > 2 units/day
* Aberrations in kidney, liver and thyroid function
* Use of any experimental medication within 6 months of the study
* The use of immunosuppressive drugs

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Postprandial change in leukocyte activation | area under the curve during 2 hours
  Leukocyte activation is determined by flow cytometry, using fluorescent labelled antibodies: FITC-conjugated anti-CD66b and PE-conjugated anti-CD11b, expressed in mean fluorescence intensity in arbitrary units. The difference in postprandial response, expressed as area under the curve, between patients with T2DM, FCH and healthy controls is determined using ANOVA.

SECONDARY OUTCOMES:
Correlation between chronic glycemia and leukocyte activation | area under the curve during 2 hours
  To assess whether chronic hyperglycemia (HbA1c) correlates with postprandial leukocyte activation, correlation between HbA1c and postprandial leukocyte activation (area under the curve) will be determined for the total study group.
Correlation between acute glycemia and leukocyte activation | area under the curve during 2 hours
  To assess whether acute hyperglycemia correlates with postprandial leukocyte activation, correlation between fasting glucose levels and postprandial leukocyte activation (area under the curve) will be determined for the total study group.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Castro Cabezas, MD, PhD, Study Chair — Sint Franciscus Gasthuis

REFERENCES:
- [Derived] de Vries MA, Alipour A, Klop B, van de Geijn GJ, Janssen HW, Njo TL, van der Meulen N, Rietveld AP, Liem AH, Westerman EM, de Herder WW, Cabezas MC. Glucose-dependent leukocyte activation in patients with type 2 diabetes mellitus, familial combined hyperlipidemia and healthy controls. Metabolism. 2015 Feb;64(2):213-7. doi: 10.1016/j.metabol.2014.10.011. Epub 2014 Oct 16. PMID 25456098